CLINICAL TRIAL: NCT03107026
Title: A 12-week, Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-dosed, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Dasotraline in Adults With Moderate to Severe Binge Eating Disorder
Brief Title: A Study to Evaluate a Drug (Dasotraline) on the Safety, Effectiveness and How Well the Body Tolerates it, in Adults With Moderate to Severe Binge Eating Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP360-321
Record Dates: First submitted 2017-03-17; First posted 2017-04-11 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Binge Eating Disorder
Keywords: Binge eating Disorder; dasotraline
MeSH Terms: conditions — Binge-Eating Disorder | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine; SEP 225289

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dasotraline 4mg (Experimental): dasotraline 4mg once daily
  Interventions: Drug: dasotraline 4mg
- dasotraline 6mg (Experimental): dasotraline 6mg once daily
  Interventions: Drug: dasotraline 6mg
- Placebo (Placebo Comparator): Placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dasotraline 4mg — dasotraline 4mg tablet once daily
  Other Names: SEP225289
  Arms: dasotraline 4mg
Drug: dasotraline 6mg — dasotraline 6mg tablet once daily
  Other Names: SEP225289
  Arms: dasotraline 6mg
Drug: Placebo — Placebo tablet once daily
  Arms: Placebo

SUMMARY:
A study to evaluate a drug (dasotraline) on the safety, effectiveness and how well the body tolerates it, in adults with moderate to severe binge eating disorder

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, multicenter, outpatient study evaluating the efficacy and safety of 2 doses of dasotraline (4 and 6 mg/day) versus placebo over a 12-week treatment period in adults with BED. This study is projected to randomize approximately 480 subjects to 3 treatment groups in a 1:1:1 ratio (4 mg/day dasotraline, 6 mg/day dasotraline, and placebo).

Subjects randomized to placebo will receive placebo for the duration of the treatment period.

Subjects randomized to 4 mg/day dasotraline will receive 4 mg/day for the duration of the treatment period.

Subjects randomized to 6 mg/day dasotraline will be dosed with 4 mg/day dasotraline for the first 2 weeks of the treatment period and will be increased to 6 mg/day at Week 2.

If, in the judgment of the Investigator, the subject does not tolerate the assigned dose, he or she will be discontinued from the study.

The study will consist of 3 periods: Screening (up to 3 weeks), 12-weeks of treatment, and a 3-week study drug withdrawal period. Subjects who complete the 12-week double-blind treatment period in this study may be eligible to enroll and continue treatment for an additional 12 months in an open-label extension study (Study SEP360-322). Subjects who do not enter the extension study will complete the study drug withdrawal period in this study.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female subject between 18-55 years of age, inclusive, at time of informed consent.

2. Subject meets the following DSM-5 criteria for a diagnosis of BED. An episode of binge eating is characterized by both:

* Eating an amount of food larger than what most people would eat, in a discrete period of time (eg, 2 hours)
* Sense of lack of control over eating episode

Binge eating episodes are associated with ≥ 3 of the following:

* Eating much more rapidly than normal
* Eating until uncomfortably full
* Eating large amounts when not feeling hungry
* Eating alone because of embarrassment
* Feeling disgusted with oneself, guilty afterward Binge eating episodes are also associated with marked distress regarding the episode and not associated with recurrent use of compensatory behavior (eg, bulimia nervosa). Note: A subject using compensatory behavior less than 1 time every 2 weeks over the 3 months prior to screening may be permitted to enroll in the study.

  3. Diagnosis is confirmed based on the Structured Clinical Interview for DSM-IV Axis I Disorders, Module H (SCID-I Module H), clinician review of subject diaries, and the EDE-Q.

  4. Subject has a BED diagnosis or is diagnosed at screening and has a history of at least 2 binge eating days a week for at least 6 months prior to screening.

  5. Subject's BED is of at least moderate severity with subject reporting at least 3 binge eating days for each of the 2 weeks prior to baseline as documented in the subject's binge diary. A binge eating day is defined as having at least one binge eating episode 6. Subject has a BE- CGI-S score ≥ 4 at screening and baseline. 7. Subject has a negative breath alcohol test and a negative UDS for any illicit drug.

  8. Female subject must have a negative serum pregnancy test at screening; females who are post-menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.

  9. Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to use an effective and medically acceptable form of birth control throughout the study period. Note: Continued use of an effective and medically acceptable form of birth control is recommended for 30 days after study completion.

  10. Subject must be able to comply with study drug administration and adhere to protocol requirements including all study assessments.

  11. Subject can read well enough to understand the informed consent form and other subject materials

Exclusion Criteria:

1. Subject has BMI of 18 kg/m2or less, or greater than 45 kg/m2.
2. Subject has a lifetime history or current symptoms consistent with bulimia nervosa or anorexia nervosa.
3. Subject has started psychotherapy (eg, supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) within 3 months prior to screening. Note: Subjects receiving stable ongoing psychotherapy for longer than 3 months are permitted to enroll.
4. Subject has participated in a formal weight loss program (eg, Weight Watchers®) within 3 months prior to screening.
5. Subject has used a psychostimulant or mood stabilizer within the 3 months prior to screening.
6. Subject has used any medications for the treatment of binge eating, other eating disorders, obesity, or weight gain or any other medication that could result in weight gain or weight loss including over-the-counter and herbal products within the 3 months prior to screening.
7. Subject has received lisdexamfetamine dimesylate (Vyvanse®) for any reason, including but not limited to participation in any Phase 2 or 3 trial.
8. Subject has a lifetime history of psychotic disorder, bipolar disorder, hypomania, dementia, or ADHD as defined by the DSM-5 criteria.
9. Subject has a history of moderate to severe depression based on Investigator's judgment within the 6 months prior to screening or is currently taking or has taken any medication for depression during the 3 months prior to screening.
10. Subject has MADRS score ≥ 18 at screening and Baseline visit.
11. Subject has a history of substance use disorder including alcohol use disorder (excluding nicotine and caffeine) within the 12 months prior to screening, as defined by the DSM-5 criteria.
12. Subject is considered a suicide risk in the investigator's opinion or has any previous history of suicide attempt within the past 12 months.
13. Subject answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at screening (in the past month). Subjects who answer "yes" to this question must be referred to the Investigator for follow-up evaluation.
14. Subject has type I diabetes mellitus or insulin-dependent diabetes mellitus.
15. Subject with type II diabetes mellitus, has hemoglobin A1c ≥ 6.5% at screening, or has initiated treatment with or changed the dose of a glucose-lowering agent within 3 months prior to screening.
16. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, documented heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
17. Subject has initiated treatment with or changed the dose of a lipid-lowering medication within the 3 months prior to screening.
18. Subject has a history of moderate or severe hypertension that in the Investigator's opinion has not been medically stable or has required a change in dosage and/or medication during the 3 months prior to screening.
19. Subject has a history of focal or diffuse brain disorder including but not limited to epilepsy, seizures (except childhood febrile seizures),stroke, benign or malignant tumors, or head trauma with loss of consciousness lasting more than 5 minutes; unexplained syncope or other unexplained blackouts (except single incident); or a history of clinically significant repeated head-traumas without loss of consciousness.
20. Subject has had polycystic ovarian syndrome (PCOS) in the previous 12 months, even if no treatment was provided.
21. Subject is female and pregnant or nursing.
22. Subject has had major bariatric surgery, eg, gastric jejunal bypass,Roux-en-Y gastric bypass, sleeve gastrectomy, duodenal switch with biliopancreatic diversion for weight loss at any time.
23. Minor bariatric surgey (eg, lap bands) within 3 years of screening. Note: Surgeries for cosmetic reasons are not exclusionary but should be discussed with the medical monitor.
24. Subject has a history of positive test for either Hepatitis B surface antigen or Hepatitis C antibody, and has liver function test results at screening above the upper limit of normal (ULN) for the reference laboratory.
25. Subject without a history of positive test for Hepatitis B surface antigen or Hepatitis C antibody has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the ULN at screening.
26. Subject has a blood urea nitrogen (BUN) value ≥ 1.5 times the ULN for the reference range, serum creatinine > 1.5 times the ULN for the reference range, fasting blood glucose ≥ 126 mg/dL (7.0 mmol/L), or hemoglobin A1c ≥ 6.5% at screening.
27. Subject is known to have tested positive for human immunodeficiency virus (HIV).
28. Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, ECG, or laboratory tests that the Investigator considers to be inappropriate to allow participation in the study.
29. The subject's screening ECG shows a corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec for male subjects or ≥ 470 msec for female subjects. Eligibility will be based on the core laboratory ECG interpretation report.
30. Subject has any life-time history of abuse or diversion of stimulants.
31. Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
32. Subject who in the opinion of the Sponsor and Investigator has any other psychiatric or medical condition or disorder or any other psychosocial or work-related issue not previously listed that could interfere with the diagnosis of BED at screening or subsequent evaluations during the course of the study.
33. Subject who may experience or who is currently experiencing significant psychosocial or environmental stressors (eg, loss of employment, loss of housing, financial hardship, divorce) that could impede their ability to adhere to protocol requirements, as judged by the Investigator.
34. Subject is currently participating in or has participated in any clinical trial within the last 90 days or has participated in more than 2 clinical trials within the past year. This includes studies using marketed compounds or devices.
35. Subject has previously been enrolled in a clinical trial of dasotraline (SEP-225289).
36. Subject is an investigational site staff member or the relative of an investigational site staff member.
37. Subject has started a new physical training/exercise program for the purpose of managing his or her weight or binge eating within 3 months prior to screening. Note: Subjects participating in a stable physical training/exercise program for longer than 3 months are permitted to enroll.
38. Subject has a history of malignancy within 5 years prior to the Screening visit, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. History of pituitary tumor, whether benign or malignant, is exclusionary.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 491 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (50):
- United States (50):
  - NoesisPharma, LLC, Phoenix, Arizona
  - Southern California Research, Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative NeuroScience Network, LLC, Garden Grove, California
  - Pharmacology Research Institute, Newport Beach, California
  - PCSD- Feighner Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Syrentis Clinical Research, Santa Ana, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Lytle and Weiss PLLC, Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Miami Research Associates, South Miami, Florida
  - Institute for Advanced Medical Research at Mercer University, Atlanta, Georgia
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Northwest ehavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Prairie Health and Wellness, Wichita, Kansas
  - McLean Hospital Harvard Medical School, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Inc, Methuen, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Rocheser Center for Behavioral Medicine, Rochester Hills, Michigan
  - Midwest Research Group - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - ActivMed Practice and Research, Inc, Portsmouth, New Hampshire
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Manhattan Behavior Medicine, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radient Research, Akron, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Linder Center of Hope, Mason, Ohio
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Costal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Donald J. Garcia, MD, PA, Austin, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 491 subjects were randomized in this study. Five subjects were randomized but never received any dose of study medication.
Period: Overall Study
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Started | 163 | 161 | 162
Completed | 131 | 123 | 106
Not Completed | 32 | 38 | 56
Not completed — Adverse Event | 2 | 14 | 23
Not completed — Lost to Follow-up | 12 | 12 | 13
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 5 | 17
Not completed — non compliance with study visits | 1 | 2 | 0
Not completed — non-compliance with study drug | 2 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg | Total
Number analyzed (Participants) | 163 | 161 | 162 | 486
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 4
  Between 18 and 65 years | 162 | 160 | 160 | 482
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (10.26) | 36.9 (9.55) | 38.9 (9.7) | 37.7 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 138 | 133 | 408
  Male | 26 | 23 | 29 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 31 | 26 | 85
  Not Hispanic or Latino | 135 | 130 | 136 | 401
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 1 | 7 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 29 | 25 | 32 | 86
  White | 131 | 119 | 121 | 371
  More than one race | 2 | 8 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 167.4 (8.64) | 166.8 (8.33) | 167.3 (8.22) | 167.2 (8.38)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 96.9 (20.79) | 96.9 (19.69) | 96.1 (17.97) | 96.6 (19.48)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.46 (6.283) | 34.76 (6.073) | 34.27 (5.743) | 34.5 (6.028)
Number of Binge Eating Days per Week at Baseline [Mean (Standard Deviation); unit: binge eating days/week] | 4.26 (0.994) | 4.22 (1.115) | 4.19 (1.069) | 4.22 (1.058)
Binge-eating Clinical Global Impression-Severity (BE-CGI-S) score at Baseline [Mean (Standard Deviation); unit: units on a scale] | 4.4 (0.51) | 4.5 (0.51) | 4.4 (0.51) | 4.4 (0.51)
Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) total score at Baseline [Mean (Standard Deviation); unit: units on a scale] | 21.9 (3.66) | 21.6 (3.71) | 21.6 (4.29) | 21.7 (3.89)
BMI category [Count of Participants; unit: Participants]
  Underweight/Normal (<25) | 12 | 9 | 8 | 29
  Overweight (25 to <30) | 28 | 32 | 30 | 90
  Obesity Class I (30 to <35) | 43 | 41 | 48 | 132
  Obesity Class II (35 to <40) | 46 | 46 | 45 | 137
  Obesity Class III (>=40) | 34 | 33 | 31 | 98
Number of Binge Eating Episodes per Week at Baseline [Mean (Standard Deviation); unit: Binge eating episodes/week] | 5.59 (2.803) | 5.42 (3.546) | 5.35 (2.992) | 5.45 (3.123)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Binge Days
Description: Change from baseline in number of binge days (defined as days during which at least 1 binge episode occurs) per week at Week 12
Time Frame: baseline and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: binge days/week
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
binge days/week | -2.92 (0.134) | -3.21 (0.135) | -3.47 (0.140)
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Test type: Superiority; p = 0.1187, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.66 to 0.08], Standard Error of Mean 0.187
Statistical Analysis 2: Comparison: Placebo vs Dasotraline 6mg; Test type: Superiority; p = 0.0045, Mixed Models Analysis; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.93 to -0.17], Standard Error of Mean 0.192

2. Secondary Outcome: Change From Baseline in Binge Eating Clinical Global Impression-Severity( BE-CGI-S )Score
Description: Binge-eating Clinical Global Impression-Severity (BE-CGI-S) The BE-CGI-S is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
Time Frame: baseline and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale | -1.77 (0.114) | -2.13 (0.117) | -2.27 (0.121)
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Test type: Superiority; p = 0.0256, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.68 to -0.04], Standard Error of Mean 0.162
Statistical Analysis 2: Comparison: Placebo vs Dasotraline 6mg; Test type: Superiority; p = 0.0025, Mixed Models Analysis; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-0.83 to -0.18], Standard Error of Mean 0.166

3. Secondary Outcome: Percent of Subjects With a 4-week Cessation From Binge Eating
Description: Percent of subjects with a 4-week cessation from binge eating (defined as a 100% reduction for at least 28 consecutive days in the number of binge eating episodes prior to Week 12/end of treatment [EOT])
Time Frame: up to 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
Participants | 49 | 54 | 55
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Test type: Superiority; p = 0.5342, Regression, Logistic; Odds Ratio (OR) = 1.160, 95% CI 2-sided [0.726 to 1.854]
Statistical Analysis 2: Comparison: Placebo vs Dasotraline 6mg; Test type: Superiority; p = 0.4905, Regression, Logistic; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.738 to 1.882]

4. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Total Score
Description: Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Y-BOCS-BE total scores range from 0 to 40. Y-BOCS-BE obsessions subscale ranges from 0 to 20. Y-BOCS-BE compulsions subscale ranges from 0 to 20. Higher values of Y-BOCS-BE score and subscale scores represent greater severity of illness
Time Frame: baseline and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale | -11.83 (0.670) | -14.13 (0.680) | -15.23 (0.703)
Statistical Analysis 1: Comparison: Placebo vs Dasotraline 4mg; Test type: Superiority; p = 0.0154, Mixed Models Analysis; Mean Difference (Final Values) = -2.30, 95% CI 2-sided [-4.16 to -0.44], Standard Error of Mean 0.946
Statistical Analysis 2: Comparison: Placebo vs Dasotraline 6mg; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Mean Difference (Net) = -3.40, 95% CI 2-sided [-5.31 to -1.50], Standard Error of Mean 0.969

5. Secondary Outcome: Change From Baseline in Number of Binge Days Per Week at Weeks 1, 2, 3, 4, 6, 8, and 10
Description: Change from baseline in number of binge days per week at Weeks 1, 2, 3, 4, 6, 8, and 10
Time Frame: baseline and up to 10 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: binge days/week
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
binge days/week
  Week 1 | -1.16 (0.137) | -1.82 (0.137) | -1.51 (0.136)
  Week 2 | -1.74 (0.137) | -2.36 (0.138) | -2.27 (0.136)
  Week 3 | -2.23 (0.135) | -2.74 (0.136) | -2.70 (0.135)
  Week 4 | -2.27 (0.143) | -2.85 (0.144) | -2.98 (0.145)
  Week 6 | -2.61 (0.126) | -2.97 (0.127) | -3.24 (0.130)
  Week 8 | -2.80 (0.127) | -3.15 (0.127) | -3.31 (0.132)
  Week 10 | -2.87 (0.128) | -3.12 (0.129) | -3.31 (0.134)

6. Secondary Outcome: Change From Baseline in Number of Binge Episodes Per Week at Weeks 1, 2, 3, 4, 6, 8, 10, and 12
Description: Change from baseline in number of binge episodes per week at Weeks 1, 2, 3, 4, 6, 8, 10, and 12
Time Frame: baseline and up to 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: binge episodes
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
binge episodes
  Week 1 | -1.53 (0.230) | -2.43 (0.231) | -2.21 (0.230)
  Week 2 | -2.48 (0.235) | -3.20 (0.237) | -2.88 (0.234)
  Week 3 | -3.06 (0.226) | -3.69 (0.228) | -3.46 (0.226)
  Week 4 | -2.95 (0.254) | -3.72 (0.256) | -3.77 (0.257)
  Week 6 | -3.43 (0.231) | -3.90 (0.234) | -4.06 (0.236)
  Week 8 | -3.64 (0.216) | -4.20 (0.218) | -4.19 (0.223)
  Week 10 | -3.67 (0.213) | -4.17 (0.215) | -4.25 (0.221)
  week 12 | -3.70 (0.227) | -4.32 (0.230) | -4.38 (0.237)

7. Secondary Outcome: Change From Baseline in Binge-eating Clinical Global Impression-Severity (BE-CGI-S) Score at Weeks 2, 4, 6, 8, and 10
Description: as for outcome 2
Time Frame: baseline and up to 10 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale
  Week 2 | -0.82 (0.090) | -1.37 (0.091) | -1.20 (0.090)
  Week 4 | -1.21 (0.102) | -1.89 (0.104) | -1.79 (0.102)
  Week 6 | -1.37 (0.105) | -1.83 (0.107) | -1.90 (0.108)
  Week 8 | -1.55 (0.108) | -1.91 (0.110) | -2.04 (0.113)
  Week 10 | -1.59 (0.112) | -1.95 (0.115) | -2.07 (0.119)

8. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Total Score at Weeks 2, 4, 6, 8, and 10
Description: as for outcome 4
Time Frame: baseline and up to 10 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale
  Week 2 | -6.49 (0.576) | -10.32 (0.583) | -9.21 (0.577)
  Week 4 | -9.30 (0.623) | -13.15 (0.631) | -12.77 (0.627)
  Week 6 | -9.74 (0.645) | -12.50 (0.653) | -13.65 (0.663)
  Week 8 | -10.99 (0.654) | -13.55 (0.661) | -14.25 (0.681)
  Week 10 | -10.81 (0.658) | -13.54 (0.668) | -14.21 (0.690)

9. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y-BOCS-BE) Subscale Scores (Obsessions and Compulsions) at Weeks 2, 4, 6, 8, 10, and 12
Description: as for outcome 4
Time Frame: baseline and up to 12 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale
  Obsessions Subscale Score Week 2 | -3.14 (0.297) | -4.84 (0.301) | -4.37 (0.297)
  Obsessions Subscale Score Week 4 | -4.30 (0.315) | -6.32 (0.319) | -6.29 (0.317)
  Obsessions Subscale Score Week 6 | -4.65 (0.326) | -6.12 (0.330) | -6.70 (0.336)
  Obsessions Subscale Score Week 8 | -5.20 (0.337) | -6.48 (0.341) | -7.00 (0.354)
  Obsessions Subscale Score Week 10 | -4.94 (0.335) | -6.49 (0.340) | -6.88 (0.353)
  Obsessions Subscale Score Week 12 | -5.56 (0.339) | -6.73 (0.344) | -7.43 (0.356)
  Compulsions Subscale Score Week 2 | -3.32 (0.303) | -5.45 (0.307) | -4.83 (0.304)
  Compulsions Subscale Score Week 4 | -4.98 (0.330) | -6.80 (0.334) | -6.44 (0.333)
  Compulsions Subscale Score Week 6 | -5.08 (0.337) | -6.34 (0.341) | -6.91 (0.348)
  Compulsions Subscale Score Week 8 | -5.77 (0.343) | -7.03 (0.347) | -7.22 (0.359)
  Compulsions Subscale Score Week 10 | -5.85 (0.344) | -7.00 (0.349) | -7.30 (0.361)
  Compulsions Subscale Score Week 12 | -6.24 (0.352) | -7.34 (0.357) | -7.78 (0.370)

10. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score and Subscale Scores (School/Work Disability, Social Life Disability, and Family Life Disability) at Weeks 6 and 12
Description: Sheehan Disability Scale (SDS) total and subscale scores The Sheehan Disability Scale (SDS) 3 subscales (work/school, social life, home life) are rated on the following scale: 0 = not at all; 1-3 = mildly; 4-6 = moderately; 7-9 =markedly; 10 = extremely. The 3 items can be combined into a single global measure of impairment (SDS total score) that ranges from 0 (unimpaired) to 30 (highly impaired). A higher subscale score and total score are associated with greater illness severity
Time Frame: baseline and 6 Weeks and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale
  SDS Total Score Week 6 | -5.73 (0.551) | -7.65 (0.563) | -6.88 (0.566)
  SDS Total Score Week 12 | -6.14 (0.547) | -8.56 (0.551) | -8.19 (0.580)
  SDS Work/School Week 6 | -1.20 (0.185) | -1.81 (0.189) | -1.57 (0.191)
  SDS Work/School Week 12 | -1.33 (0.189) | -1.93 (0.190) | -1.84 (0.201)
  SDS Social Life Week 6 | -2.26 (0.199) | -3.06 (0.199) | -2.82 (0.203)
  SDS Social Life Week 12 | -2.38 (0.195) | -3.50 (0.196) | -3.38 (0.207)
  SDS Family Life/Home Responsibilities Week 6 | -2.04 (0.188) | -2.59 (0.188) | -2.40 (0.192)
  SDS Family Life/Home Responsibilities Week 12 | -2.39 (0.177) | -2.94 (0.178) | -3.00 (0.189)

11. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 12
Description: Montgomery-Asberg Depression Rating Scale (MADRS) total score The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
Time Frame: baseline and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale | -1.1 (0.36) | -0.9 (0.36) | 0.6 (0.36)

12. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Week 12
Description: Hamilton Anxiety Rating Scale (HAM-A) total score HAM-A total score ranges from 0 to 56. A higher score is associated with a greater degree of anxiety.
Time Frame: baseline and 12 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale | -0.4 (0.37) | 0.3 (0.37) | 1.8 (0.37)

13. Secondary Outcome: Proportion of Binge Eating Responders Who Have ≥ 75% Reduction in the Number of Binge Eating Episodes From Baseline at Week 12
Description: Proportion of binge eating responders who have ≥ 75% reduction in the number of binge eating episodes from Baseline at Week 12
Time Frame: 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
Participants | 91 | 112 | 123

14. Secondary Outcome: Change From Baseline in Eating Disorder Examination Questionnaire (EDE-Q) Modified Including EDE-Q7 Global Score and 3 Subscale Scores (Dietary Restraint, Shape/Weight Overvaluation, and Body Dissatisfaction) at Week 12
Description: Eating Disorder Examination Questionnaire (EDE-Q) Modified global and subscale scores 4 subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) range from 0- 6, where 0 represents absence of the feature and 6 represents an extreme degree. An EDE-Q global score is calculated as average of 4 EDE-Q subscale scores.
Time Frame: baseline and 2 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
Number analyzed (Participants) | 162 | 161 | 162
units on a scale
  EDE-QM Global Score Week 12 LOCF | -0.54 (0.116) | -1.20 (0.116) | -1.35 (0.118)
  EDE-QM Restraint Week 12 LOCF | -0.23 (0.149) | -0.85 (0.149) | -1.14 (0.152)
  EDE-QM Shape Concern Week 12 LOCF | -0.74 (0.132) | -1.36 (0.132) | -1.43 (0.135)
  EDE-QM Weight Concern Week 12 LOCF | -0.62 (0.129) | -1.38 (0.130) | -1.46 (0.132)

ADVERSE EVENTS:
Time Frame: An AE with a start date on or after the date of first dose through 7 days after study drug discontinuation (14 days for serious adverse events and deaths) for subjects who complete or discontinue this study but do not enter into the extension study), or through the last study day of the double-blind treatment period for subjects continuing into the extension study (double-blind treatment duration: 12 weeks)
Description: An AE with a start date on or after the date of first dose through 7 days after study drug discontinuation (14 days for serious adverse events and deaths) for subjects who complete or discontinue this study but do not enter into the extension study), or through the last study day of the double-blind treatment period for subjects continuing into the extension study (double-blind treatment duration: 12 weeks)
Arm/Group | Placebo | Dasotraline 4mg | Dasotraline 6mg
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/161 | 0/162
Serious Adverse Events (participants affected / at risk) | 1/163 | 3/161 | 1/162
Other Adverse Events (participants affected / at risk) | 70/163 | 105/161 | 113/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=163) | Dasotraline 4mg (N=161) | Dasotraline 6mg (N=162)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=163) | Dasotraline 4mg (N=161) | Dasotraline 6mg (N=162)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (6) | 11 (11)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 34 (34) | 43 (45)
Nausea (Gastrointestinal disorders) | 9 (10) | 19 (22) | 21 (25)
Upper respiratory tract infection (Infections and infestations) | 23 (25) | 11 (13) | 13 (14)
Weight decreased (Investigations) | 2 (2) | 14 (14) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 15 (15) | 26 (28)
Dizziness (Nervous system disorders) | 3 (3) | 8 (8) | 9 (9)
Headache (Nervous system disorders) | 17 (18) | 20 (23) | 27 (29)
Anxiety (Psychiatric disorders) | 4 (4) | 14 (14) | 22 (24)
Initial insomnia (Psychiatric disorders) | 4 (5) | 10 (10) | 14 (15)
Insomnia (Psychiatric disorders) | 17 (17) | 34 (35) | 45 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03107026/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03107026/SAP_001.pdf